CLINICAL TRIAL: NCT06579027
Title: A Novel, Child-friendly, Home-based Navigation Training Program Using Joystick-operated Ride-on Toys to Improve Upper Extremity Function in Children With Hemiplegia: A Pilot Study
Brief Title: A Novel Program Using Ride-on Toys to Improve Upper Extremity Function in Children With Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sudha Srinivasan, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-10-800-910; 1R21HD109605-01A1 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hemiplegia; Cerebral Palsy; Children, Only
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SPEED (Strength and Power in upper Extremities through Exploratory Driving) (Experimental): Children will receive training focused on improving affected arm function using modified, joystick-operated ride-on toys. The commercial ride-on toys will be modified to allow operation in a single joystick control mode provided on the child's affected side. The manualized SPEED sessions will involve 2 components: (a) Multidirectional navigational games where children will use their affected UE to drive and maneuver the toy and (b) Object-based UE tasks completed at intermediate stops/stations during navigation. Navigational opportunities will encourage children to navigate through paths of different shapes, sizes, and complexity levels (e.g., straight, circle, diamond, slalom, obstacle courses etc.) Object-based tasks will encourage functional UE movement patterns during object interactions such as reaching, throwing, catching, pulling, pushing, lifting, knocking, holding, grasping, opening, closing, release, and manipulation.
  Interventions: Device: SPEED Training
- CRAFT (Creative Rehabilitation for Arm Functional Training) (Active Comparator): Children will engage in seated creative motor games focused on promoting gross and fine motor UE function. Training sessions will encourage use of the affected UE during unimanual and bimanual activities. Each training session will involve the following components: (a) Stretching exercises and (b) Task-oriented strengthening activities. Stretching exercises will involve range of motion exercises to encourage active warmup of proximal (shoulder, elbow) and distal (wrist, hand) UE muscles and movement dissociation. Task-oriented strengthening will involve use of the affected UE as a mobilizer and a stabilizer during building (e.g., Play-Doh, blocks, puzzles) and art-craft activities (e.g., folding, cutting, pasting, coloring). Task-oriented practice will emphasize skills such as reaching, grasping, release, and manipulation of training supplies.
  Interventions: Behavioral: CRAFT Training

INTERVENTIONS:
Device: SPEED Training — Children will use ride-on toys controlled using their affected arm to navigate through their environment and complete playful theme-based challenges. Children will use their affected UE during navigation to start and stop the toy, move steadily forward and backward, turn to the right and left, perform 180° and 360° turns to either side, and avoid obstacles. Children will complete object-based UE tasks requiring gross and fine motor control at intermediate stops during navigation. Navigational tasks will be progressed by increasing complexity of paths (straight to slalom paths needing more directional changes), spaces (wide to narrow spaces), and precision (obstacle courses and mazes requiring skillful navigation, motor planning, and route finding). Object-based tasks will be progressed in terms of force requirements (small to large forces), range of motion (near to far reaches), precision (manipulation of large to small objects), and speed of movements (slow to fast).
  Other Names: Strength and Power in upper Extremities through Exploratory Driving
  Arms: SPEED (Strength and Power in upper Extremities through Exploratory Driving)
Behavioral: CRAFT Training — Children will engage in predominantly seated activities based on conventional occupational therapy to promote unimanual and bimanual UE function. Training sessions will be based on playful child-friendly themes (e.g., dinosaurs, space exploration, aquatic theme, etc.) and all training activities will incorporate the session theme. Activities will involve practice of functional gross and fine motor UE movement patterns that children typically use during daily life. Training will emphasize the use of the affected UE in different roles (i.e., stabilizer, mobilizer, and active and passive assist) during warm-up, building, and art-craft activities. The training will be progressed in terms of forces needed, range of motion, precision, and movement speed.
  Other Names: Creative Rehabilitation for Arm Functional Training
  Arms: CRAFT (Creative Rehabilitation for Arm Functional Training)

SUMMARY:
The purpose of this study is to assess the feasibility and utility of 2 types of play-based training programs co-delivered by researchers and caregivers within home/community settings to promote arm function among 3-to-8-year-old children with hemiplegia. Specifically, investigators will assess the feasibility of implementation and acceptance/satisfaction associated with a researcher-caregiver co-delivered community-based training program involving either joystick-operated powered ride-on toys (SPEED training) or creative upper extremity training (CRAFT training).

The investigators will also compare the effects of these 2 types of training programs on children's arm motor function and spontaneous use of their affected arm during daily activities.

DETAILED DESCRIPTION:
Prior to the start of the study, researchers will conduct a phone screening with the family to confirm their child's eligibility to participate in the study. Once eligibility is confirmed, during the pretest session (week 1), standardized assessments will be conducted to evaluate the child's ability to use their affected arm for different functional activities. During this testing visit, researchers will also attach small sensors on the child's arms and ask them to complete arm movements and functional tasks (e.g., lifting blocks and putting them into a small cup). At the pretest, the child will also be provided 2 activity monitors (similar to wrist watches) to wear on both wrists for 1 week. The activity monitors will allow the researchers to track the child's habitual arm activity over the duration of a week. In addition, caregivers will be asked to complete questionnaires to obtain information on their child's overall health, development, and their ability to use their affected arm for various activities of daily living.

Assessments and questionnaires will be repeated again at the posttest (i.e., at week 8 that corresponds with completion of the 6-week intervention phase) and at 1-month follow-up following intervention completion (i.e., week 12).

Following the pretest, the child will be randomized into one of the training groups (SPEED or CRAFT). During the 6-week intervention phase, the research team will visit the child's home/community 2 times/week to provide the training. Caregivers will be requested to practice 2 additional sessions every week with their child in both groups.

Children in the Strength and Power in upper Extremities through Exploratory Driving (SPEED) training group will engage in multidirectional navigation games and object-based upper extremity quests using the ride-on toys. The toy will be modified to enable operation in a single joystick control mode with the joystick control provided on the child's affected side. The training activities will be designed to encourage children to use their affected arm for training activities. The training will involve children driving through incrementally challenging courses/paths and completing object-based tasks that require use of their affected arm for reaching, grasping, release, and fine manipulation activities. Children will be asked to wear a mitten on their unaffected hand during the sessions. Children in the Creative Rehabilitation for Arm Functional Training (CRAFT) group will engage in seated creative motor games that will encourage use of their affected arm. Training activities will involve stretching and strengthening exercises, building activities (e.g., using Play-doh, blocks, etc.), and art-craft projects, all of which will require the skillful use of the affected arm for reach, grasp, release, and manipulation activities.

Research-delivered sessions in both groups will last around 30-45 minutes. Caregivers will be encouraged to provide 2 more sessions every week lasting about 15-20 minutes/session. The research team will provide caregivers in both groups with the required materials for caregiver sessions. In the SPEED group, the ride-on toy will be left with the family for the duration of the intervention (i.e., 6 weeks). Both researchers and caregivers will be asked to keep track of training sessions (duration, frequency, etc.) using a training log. During the course of the study, children in both groups will continue to receive treatment-as-usual through school or private settings. Families will be asked to log the therapies their child is receiving every week over the course of the study using a training diary (# of times/week, duration of each session, type of therapy received) provided by the researchers. Researchers will video record all testing and researcher-delivered training sessions so that children's performance can be scored later.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between the ages of 3 - 8 years
* Diagnosed with hemiplegia by a medical doctor with clear asymmetry in upper extremity strength and control (i.e., one upper limb is clearly weaker than the other)
* Can maintain a supported sitting position for at least 15 minutes

Exclusion Criteria:

* Only lower limb involvement
* Recent history (within past 6 months) of trauma or surgery or Botox
* Uncorrected blindness/profound visual impairment
* Fixed deformities at wrist or hand
* No active control in affected UE
* Inability to follow 2-step directions
* Weight > 150 lbs.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence | From start to end of the 6-week intervention phase on a weekly basis
  Researchers and caregivers will maintain training logs to document the frequency (# of sessions/week) and duration (time per session) of training sessions. In the SPEED group, the ride-on toy will collect data on amount of device use during training sessions.
Treatment retention | From date of randomization to date of the final data collection visit with the last participant, assessed over 24 months
  Researchers will report treatment retention (# of families who withdrew). The researchers will track the # of families who withdrew from the study, the timepoint within the study timeline of withdrawal, and the reasons for withdrawal.
Treatment satisfaction | At 8 weeks (i.e., at the posttest visit conducted following completion of the 6-week intervention phase)
  The researchers will use the 16-item Physical Activity Enjoyment Scale (PAES) with children (delivered in an interview format) scored on a Likert scale of 1 (Disagree a lot) to 5 (Agree a lot) at posttest to assess perceived competence, pleasure/enjoyment, control, and sense of success. Caregivers will complete exit questionnaires/interviews to assess perceived program satisfaction, burden, willingness to continue training beyond the study, likelihood of recommending training to others, and child motivation/engagement during the training.
Changes in use of affected arm in functional activities | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of intervention phase)
  The Shriner's Hospital Upper Extremity Evaluation (SHUEE) is a video-based test that analyzes affected UE use spontaneously and on tester demand during 16 bimanual tasks in 3-18-year-olds. It has 3 components: spontaneous functional analysis (SFA), dynamic positional analysis (DPA), and grasp-release analysis (GRA), scored on a 2- to 6-point ordinal scale. The SHUEE assessment includes evaluation of spontaneous use of the involved UE and segmental alignment of the affected UE during performance of tasks on demand, for example, unscrewing a bottle cap, removing money from a wallet, putting socks on, etc. The SFA is scored on a scale from 0 to 5 where higher ratings indicate better performance. The DPA is scored on a scale from 0 to 3, where higher ratings indicate better performance. The GRA is scored on scale from 0 to 1, where higher ratings indicate better performance.
Changes in hand grip strength | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of the intervention phase)
  A calibrated digital Jamar dynamometer will be used to measure grip strength while seated with forearm supported. Following a single sub-maximal practice trial, a single maximal trial of 3-4 seconds will be collected from each hand.

SECONDARY OUTCOMES:
Changes in implementation fidelity during training sessions and factors impacting training delivery | Early (week 1), Mid (week 3), and late (week 6) training sessions within the 6-week intervention phase and at week 8 (posttest following completion of the intervention phase)
  In both training groups, a coder naïve to study aims will randomly choose and code videos (one each of early, mid, and late researcher-delivered sessions) using custom-designed fidelity checklists to assess adherence to the manualized training protocols. Caregivers will fill exit questionnaires at posttest to report ease of implementation of the training programs, barriers and facilitators related to session delivery, and adequacy of researcher support to deliver caregiver sessions.
Changes in child engagement during training sessions | Early (week 1), Mid (week 3), and Late (week 6) training sessions within the 6-week intervention phase
  The researchers will code 1 early, 1 mid, and 1 late researcher-administered session during the intervention phase in both groups (using Datavyu video coding software) to assess the child's affect and attention to the task. Specifically, in terms of affect, for each training session (early, mid, and late), researchers will code the percent duration of session spent in positive and negative affective states. In addition, training sessions (early, mid, and late session) will be coded for the child's attention patterns. The research team will code the percent duration of the session that the child attended towards task-appropriate and task-inappropriate targets. Specifically, investigators will code for attention directed towards: (a) task, (b) social partners, and (d) elsewhere.
Changes in parent-rated scores on functional use of the affected arm | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of intervention phase)
  The ABILHAND-Kids is a valid and reliable parent-rated questionnaire assessing parent perceptions of their child's level of ease or difficulty in performing 21 manual activities independently over the last 3 months. The 21 manual activities are rated by parents on a 3-point scale of "impossible", "difficult", or "easy". Items become increasingly difficult in terms of required bimanual function. Investigators will report changes in logit scores over the course of the training program.
Change in affected arm movement control | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of intervention phase)
  The Quality of Upper Extremity Skills Test (QUEST) is a criterion-referenced, valid, and reliable measure for use between 18 months-12 years to assesses quality of UE function in 4 domains: dissociated movements, grasp, protective extension, and weight bearing. The tool includes 36 items that evaluate movement patterns and hand function in children with Cerebral Palsy and are scored on a dichotomous scale (minimum value = 1, maximum value = 2), with higher scores indicating better performance. The research team will report total scores and 4 sub-domain scores on the QUEST.
Changes in independent navigational control | Early (week 1), Mid (week 3), and Late (week 6) training sessions within the 6-week intervention phase
  Early, mid, & late training sessions (one session at each time point) of children in the SPEED group will be coded for percent duration of session engaged in assisted (child needs trainer-provided manual assistance) versus independent (child is able to drive the toy unassisted) navigation.
Changes in habitual arm activity and arm asymmetry | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of intervention phase)
  Children will be asked to wear 2 wrist activity monitors (ActiGraph devices), one each on both wrists, for the duration of 1 week, at 3 time points : (a) baseline/pretest, (b) posttest following completion of the 6-week intervention phase, and (c) followup (i.e., 1 month following intervention completion). Children will be asked to wear the monitors for a period of 1 week at all 3 time points. Children will be asked to wear the monitors continuously when awake and while sleeping (minimum of 4 days - 1 weekend day and 3 weekdays) over the course of the week. Investigators will report extent of asymmetry in affected versus unaffected arm use across the time points.
Changes in maximum UE joint angles and overall range of motion on the affected arm | Baseline (i.e., pretest conducted in week 1), at 8 weeks (i.e., at posttest after completion of the 6-week intervention), and at 12 weeks (i.e., at 1-month followup after the end of intervention phase)
  Movement kinematics will be collected from both UEs during the following tasks: (a) range of motion tasks involving shoulder, elbow, forearm, and wrist movements (adapted from tasks from the QUEST and SHUEE tests) and (b) sequential bimanual tasks adapted from motor tests (i.e., clean-up task with 6 blocks requiring the child to grasp each block, transfer to the other hand, and release into a small cup). Sensors (Inertial Measurement Units (IMUs)) will be placed on both hands, both forearms, both arms, and the C7 spinous process. The research team will report maximum joint angles and overall joint range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Program, Department of Kinesiology, University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated include screening forms, participant intake forms (with demographic information, clinical information, and details of therapies received by children), parent-rated questionnaires, child-rated questionnaires, researcher-rated qualitative scales, video data from testing and training sessions, raw kinematic data, raw data from accelerometers, toy use data, training logs, and excel files generated from post-processing data collected from the study. All raw data with identifiable information will not be shared. All coded, de-identified scientific data (questionnaire responses, test scores, training logs) will be preserved and shared using Data and Specimen Hub (DASH).
Supporting Information: Study Protocol, ICF
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first.

REFERENCES:
- [Background] Srinivasan S, Amonkar N, Kumavor PD, Bubela D, Morgan K. Joystick-Operated Ride-On Toy Navigation Training for Children With Hemiplegic Cerebral Palsy: A Pilot Study. Am J Occup Ther. 2024 Jul 1;78(4):7804185070. doi: 10.5014/ajot.2024.050589. PMID 38836619
- [Background] Shahane V, Kumavor PD, Morgan K, Srinivasan S. Fast and Fun: A Pilot Feasibility Study Using Dual Joystick-Operated Ride-on Toys for Upper Extremity Rehabilitation in Children with Hemiplegia. Phys Occup Ther Pediatr. 2024;44(6):844-864. doi: 10.1080/01942638.2024.2360462. Epub 2024 Jun 11. PMID 38863174
- [Background] Srinivasan S, Kumavor PD, Morgan K. A Pilot Feasibility Study on the Use of Dual-Joystick-Operated Ride-on Toys in Upper Extremity Rehabilitation for Children with Unilateral Cerebral Palsy. Children (Basel). 2024 Mar 29;11(4):408. doi: 10.3390/children11040408. PMID 38671624
- [Background] Srinivasan S, Kumavor P, Morgan K. A Training Program Using Modified Joystick-Operated Ride-on Toys to Complement Conventional Upper Extremity Rehabilitation in Children with Cerebral Palsy: Results from a Pilot Study. Bioengineering (Basel). 2024 Mar 23;11(4):304. doi: 10.3390/bioengineering11040304. PMID 38671726
- [Background] Srinivasan S, Amonkar N, Kumavor PD, Bubela D. Measuring Upper Extremity Activity of Children With Unilateral Cerebral Palsy Using Wrist-Worn Accelerometers: A Pilot Study. Am J Occup Ther. 2024 Mar 1;78(2):7802180050. doi: 10.5014/ajot.2024.050443. PMID 38478583
- [Background] Srinivasan S, Amonkar N, Kumavor P, Morgan K, Bubela D. Outcomes Associated with a Single Joystick-Operated Ride-on-Toy Navigation Training Incorporated into a Constraint-Induced Movement Therapy Program: A Pilot Feasibility Study. Behav Sci (Basel). 2023 May 15;13(5):413. doi: 10.3390/bs13050413. PMID 37232651
- [Background] Shahane V, Kumavor P, Morgan K, Friel KM, Srinivasan SM. A protocol for a single-arm interventional study assessing the effects of a home-based joystick-operated ride-on-toy navigation training programme to improve affected upper extremity function and spontaneous use in children with unilateral cerebral palsy (UCP). BMJ Open. 2023 May 9;13(5):e071742. doi: 10.1136/bmjopen-2023-071742. PMID 37160396
- [Background] Amonkar N, Kumavor P, Morgan K, Bubela D, Srinivasan S. Feasibility of Using Joystick-Operated Ride-on-Toys to Promote Upper Extremity Function in Children With Cerebral Palsy: A Pilot Study. Pediatr Phys Ther. 2022 Oct 1;34(4):508-517. doi: 10.1097/PEP.0000000000000944. Epub 2022 Aug 30. PMID 36044637